CLINICAL TRIAL: NCT00487110
Title: Clinical Confirmation of a Pharmacodynamic Interaction Between Tropisetron and Paracetamol
Acronym: Tropisétron
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Dr Pickering Gisele, CHU Clermont-Ferrand
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU63-0021
Record Dates: First submitted 2007-06-14; First posted 2007-06-15 (Estimated); Last update posted 2010-03-29 (Estimated); Status verified 2010-03

CONDITIONS: Pain
Keywords: Pain; serotonin; interaction; Patients with postsurgical pain, after ear surgery
MeSH Terms: conditions — Pain | interventions — Tropisetron; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Tropisetron — a comparison of the analgesic action of paracetamol versus tropisetron+paracetamol
Drug: paracetamol — a comparison of the analgesic action of paracetamol versus tropisetron+paracetamol

SUMMARY:
A previous study has shown that tropisetron inhibits the analgesic effect of paracetamol in healthy volunteers. This study aims at confirming this pharmacodynamic interaction in patients with post-surgery pain.

DETAILED DESCRIPTION:
The study is a comparison of the analgesic action of paracetamol versus tropisetron + paracetamol in 30 patients who had surgery of the ear. The evaluation criteria will be the score on the visual analogue scale for pain evaluation.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years
* Men or women
* Ear surgery
* Written consent given

Exclusion Criteria:

* Paracetamol hypersensibility
* Tropisetron hypersensibility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale score will be taken at 30min, 1h, 2h, 3h and compared for the two groups | at 30 min, 1h, 2h, 3h

CONTACTS AND LOCATIONS:
Overall Officials: Pickering Gisele, MCU-PH, Principal Investigator
Locations (1):
- CHU, Clermont-Ferrand, France